CLINICAL TRIAL: NCT03888170
Title: The Impact of Pregnancy and Pregnancy-associated Hypertension on Human Uterine Myometrial Artery Reactivity
Status: Withdrawn | Type: Observational
Why Stopped: Study was never conducted
Sponsor: University of Arizona (Other)
Collaborators: Midwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: 1902347880
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy; Preeclampsia; Hypertension in Pregnancy
Keywords: Myogenic Tone; Vascular Reactivity; Vascular Remodeling
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Vascular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Blood Draw - venous blood samples will be collected from all patients for measurement of circulating hormone and inflammatory marker levels.
  2. Tissue/Amniotic Fluid Collection
     1. Samples from Cesarean section: amniotic fluid specimen, fetal membranes and placental biopsy, and a full-thickness uterine biopsy.
     2. Myometrial samples from elective hysterectomy: full-thickness uterine biopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-pregnant: Women aged 18-45 years old undergoing elective hysterectomy (either vaginal, laparoscopic, or open routes) for benign indications.
  Interventions: Other: No intervention
- Pregnant: Pregnant women aged 18-45 undergoing cesarean section at or beyond 34 weeks gestational age.
  Interventions: Other: No intervention
- Pregnant with hypertension: Pregnant women aged 18-45 undergoing cesarean section at or beyond 34 weeks gestational age with pregnancy complicate by chronic hypertension, gestational hypertension, preeclampsia without severe features, preeclampsia with severe features, or superimposed preeclampsia.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The investigators seek to describe the composition, architecture, and electrical conduction properties of the human uterine myometrial artery and their impact on vascular reactivity upon exposure to hypertensive stress. Non-pregnant women and pregnant women with and without hypertensive complications will be studied to evaluate the influence of these states on the myometrial arteries. Vascular over-reactivity and disruption of the normal pregnancy-associated physiologic changes of relaxed vascular tone possess the potential for non-compensated blood flow to the uterus and placenta that is insufficient to meet the metabolic demands of a growing placenta. With an understanding of these changes, the research team will be able to propose basic mechanistic changes of pathologic myogenic tone that may ultimately be investigated as potentially modifiable processes to reduce the development and/or severity of these pregnancy complications (gestational hypertension, preeclampsia, eclampsia, small for gestational age, intrauterine growth restriction and intrauterine fetal demise. ).

DETAILED DESCRIPTION:
The experiments proposed here seek to identify mechanisms underlying changes in the human uterine myometrial artery reactivity during pregnancy. The first series of experiments will be to address the changes that have been observed in stress-strain relationships and arterial remodeling during pregnancy. The second series of experiments will address the endothelial dependency of augmented pregnancy-induced vasoconstriction in myometrial arteries during pregnancy. Finally, the third series of experiments will be to address the unique relationship between resting membrane potential, calcium (Ca2+) signaling, and vascular reactivity in myometrial arteries from non-pregnant and pregnant women.

Blood Draw Venous blood samples will be collected from all patients for measurement of circulating hormone and inflammatory marker levels, so that vascular reactivity changes related to these components can be appropriately controlled for so as to correctly characterize similar changes attributed to either pregnancy and/or exposure to hypertensive stress.

Tissue/Amniotic Fluid Collection Samples from Cesarean section: This research protocol will include collection of the following samples at time of cesarean section - amniotic fluid specimen, fetal membranes and placental biopsy, and a full-thickness uterine biopsy specimen. There are no associated risks with collection of amniotic fluid at time of hysterotomy/amniotomy during a cesarean section or collection of the otherwise discarded placenta and fetal membranes. Generally, the risk of taking the uterine biopsy samples is no greater that of a cesarean section alone. At this time, there is no known risk of the small amount of tissue that is to be taken by biopsy. A slight increase in the incidence and magnitude of bleeding may occur. Performing these procedures under direct observation further limits this bleeding risk. Obtaining this uterine sample will add only minimal operating time and all physicians with Obstetrics & Gynecology training should be able to perform this procedure easily. A copy of the informed consent that is in place is included for review, as is a formal biopsy protocol detailing the procedure, specimen site, specimen size, storage, etc. for completing the tissue collection at time of cesarean section.

Myometrial samples from elective hysterectomy: These patients will be undergoing an elective hysterectomy that is independent of our study. Research personnel will isolate the tissue sample following surgical removal of the uterus. A copy of the informed consent that is in place for our proposed study has been included for review, as is a formal protocol documenting instructions for completing the tissue collection at time of benign, elective hysterectomy.

Laboratory Analysis Upon acquisition of collected tissue specimens, tissue will be immediately placed in containers of cold physiologic saline solution (PSS) until transport to the laboratory at Midwestern University can be arranged. Upon arrival to the laboratory, resistance-sized myometrial and placental arteries (~250 micrometers) will be dissected in cold physiologic saline solution aerated with gas containing 21% oxygen (O2), 74% nitrogen (N2), and 5% carbon dioxide (CO2).

A 1-2 mm length will be dissected, cleaned of connective tissue, and transferred to the well of a 2 mL arteriograph. The arteries are cannulated at one end, secured with suture, gently flushed free of blood and then cannulated at the distal end. The data is recorded continuously using data acquisition software (IonOptix Inc., Milton, Massachusetts, United States of America).

A pressure-servo system connected to the proximal cannula maintains a stable intraluminal pressure. Pressurized arteries are continuously superfused with physiologic saline solution (8-10 milliliters/minute) aerated with gas containing 21% O2, 74% N2 and 5% CO2 at 37 Celsius (C). After equilibration for a 120 min to obtain a stable baseline lumen diameter (LD), the myometrial artery will be constricted with 50 millimolar (mM) potassium chloride (KCl) and in the presence of 50 mM KCl, dilated with bradykinin (1 micromolar (uM)) to demonstrate intact vascular smooth muscle (VSM) and endothelial function, respectively. Vessels that do not exhibit KCl-induced constriction and/or endothelium-dependent responses will be excluded from further study. At the end of each experiment, the passive diameter of the vessel is determined by exposing the vessel to Ca2+-free PSS and diltiazem (80 mM), a L-type Ca2+-channel inhibitor.

Pressure-induced constrictions (PIC, 10 to 100mmHg) are expressed as a percent decrease of the fully dilated diameter of individual arteries at the same intravascular pressure. Diameter values will be analyzed as percent constriction or percent reversal in tone. These values will be obtained using the following equations: % constriction = [(passive diameter - active diameter) / passive diameter] X 100]; where passive represents the passive diameter of the artery in Ca2+-free PSS containing 80 mM diltiazem, and active diameter represents the diameter of the artery in response in Ca2+-containing PSS. The remaining experiments will be performed at a single intraluminal pressure of 60 millimeters of mercury (mm Hg). Whenever possible, vascular diameter will be determined simultaneously with [Ca2+] and/or intracellular electromyographic (Em) recordings.

Experimental design to assess the effect of the following inhibitors on pressure-induced constriction: L-NAME (L-nitro arginine methyl ester; to inhibit NOS), Indomethacin (INDO, to inhibit cyclooxygenase (COX)), GM6001 (to inhibit matrix metalloproteinases (MMPs)) and potassium (K+)-channel inhibitors on pressure-induced constriction. After confirming myometrial artery viability, the myometrial artery will be pressurized to 60 mm Hg, incubated for 30 minutes in the presence of one of the above inhibitors, and pressure-induced constriction (PIC) assessed. The response of the vessel in the presence of the inhibitor will be analyzed for PIC as described above and the effect of inhibitor by comparing vascular responses in its presence vs. absence.

Stress vs. strain: The contribution of elastin and collagen will be examined in myometrial artery (MA) to determine whether changes in arterial wall structure contribute to the leftward shift observed in our preliminary data. These experiments will be conducted in a manner similar to that described by Briones and colleagues. Since many of the MMPs (MMP 1, 8 and 12) act as collagenases or elastases, this will assess the contribution of MMPs on non-pregnant and pregnant MA using the non-specific MMP inhibitor, GM600157. Briefly, after obtaining control pressure curves at intraluminal pressures from 10 mmHg to 140 mmHg at 37C, in a 0 mM Ca2+ containing Krebs solution, tissues will be returned to an intraluminal pressure of 60 mmHg, re-introduced to Ca2+-containing Krebs containing elastase, collagenase or the non-specific MMP inhibitor GM6001 for 60 min, then returned to 0 mM Ca2+ containing Krebs solution plus the inhibitor for 20 min, and pressure curves will be reassessed. Pressure curves in the absence and presence of inhibitors will be compared by calculating vessel wall thickness (WT) and change wall tension (delta-T). Using the edge detection software and confirmed by histological techniques, WT will be calculated as (outer diameter - inner diameter)/2; where WT represents wall thickness (uM) and outer diameter and inner diameter represent arteriolar outer and inner diameter, respectively (micro-meter). As described by Phillips et. al.63, delta-T will be calculated as -1,333 X intraluminal pressure (PIL) X [(0.5 X Active inner diameter) - (0.5 X passive inner diameter)] X 0.0001 ; where delta-T (dynes/cm) represents the difference in wall tension between "passive" (Ca2+-free PSS) vs. "active" (Ca2+-containing PSS) conditions at a given intraluminal pressure (PIL; mmHg), and the constants 1,333 and 0.0001 are factors for converting pressure in mmHg to dynes/centimeter squared and from µm to cm, respectively. As such, delta-T represents the absolute value describing the amount by which the passive tension in the vascular wall would be increased if all active contractile mechanisms were inhibited at a given intraluminal pressure. Finally, to confirm functional studies, histological and molecular biology approaches will be employed to assess protein expression. Arterial wall thickness and wall tension will be assessed in all experiments.

Arterial wall Ca2+ measurement: To monitor changes in cytosolic Ca2+, myometrial artery will be mounted in a 2-milliliter (mL0 arteriograph and allowed to equilibrate as described above. Endothelial cell loading will be achieved by perfusing the artery intraluminally with Fura-2 (2 micro-M) and Pluronic acid (0.05%) for 5 min at room temperature. The lumen will be immediately rinsed with PSS for an additional 10 min to remove Fura-2 from the lumen and prevent vascular smooth muscle cell loading. Vascular smooth muscle cell loading will be achieved by placing Fura-2 (2 micro-M) in the vessel chamber at room temperature for 30 min. After rinsing with PSS, the vessel will be allowed to re-equilibrate for 30 min at 37 Celsius, permitting Fura-2 to de-esterify. Specificity of endothelial and smooth muscle loads will be determined using 1 micro-M bradykinin and 50 mM KCl. If the endothelium has been successfully loaded with Fura-2, bradykinin will elicit a rise in endothelial cell Ca2+ and arterial dilation. If the smooth muscle has been successfully loaded with Fura-2, bradykinin will elicit a decrease in arterial wall Ca2+ and subsequent dilation. Addition of 50 mM K+ will constrict the vessel and increase arterial wall Ca2+. The relative change in cytosolic Ca2+ will be monitored using IonOptix micro-fluorimetry equipment and changes in [Ca2+] will be calculated from the ratio of the 340 nm/380 nm excitation signal.

Electrophysiology - intracellular membrane recordings: myometrial artery segments will be cannulated similar to the method described above. Intracellular measurements will be made through the adventitial surface with micro-electrodes filled with 3 molar KCl using a Duo 773 electrometer. Successful impalements will be judged on the basis of a rapid drop in potential upon entering the cell, a low noise level and minimal change in the electrode resistance and zero potential before and after impalement. Signals will be viewed on a digital oscilloscope (Hitachi), recorded and stored for later playback using IonOptix acquisition/analysis software.

Records Review Upon participant enrollment, the medical records of each study subject will be accessed by the primary investigator. The participant will be given a study subject identification number that will be linked to the patient's medical record number only in the 'Study Participant Master List' excel spreadsheet, maintained on a password-protected, encrypted universal serial bus drive. Relevant data elements will then be reviewed and abstracted into the 'Data Collection Tool' excel spreadsheet.

Data Analysis Data analysis will be performed by the study investigators with the assistance of the Department of Biostatistics at the University of Arizona College of Medicine - Phoenix. Subject characteristics will be compared using t-tests or chi square and reported as mean ± standard error of the mean (SEM) or 95% confidence intervals as appropriate. Measurements of intrinsic vessel contractility will be compared between all subject groups under the various study conditions using t-tests, chi-square, and regression analysis where appropriate. Interim analysis will take place only when a sample size of at least 10 complete studies is obtained for each group (case and control).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years old
* Non-pregnant women undergoing elective hysterectomy (either vaginal, laparoscopic, or open routes) for benign indications.
* Pregnant women undergoing cesarean section at early-term and beyond (> 34 weeks)

Exclusion Criteria:

* Pregnancy < 34 weeks gestation.
* Non-English speaking
* Cesarean section performed with non-low transverse hysterotomy.
* History of uterine rupture or cesarean scar dehiscence, currently pregnant.
* Uterine window or significant myometrial thinning appreciated at time of surgery.
* Hysterectomy performed for treatment of malignancy
* Hysterectomy performed for risk-reduction purposes in setting of genetic predisposition to gynecologic cancer
* Diagnosis of infectious disease and/or blood borne illness
* Learning or developmental disability that precludes appropriate consenting procedures

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: Patients eligible for inclusion in this study protocol will be aged 18 years-old and older, all of which will be female. Additionally, study subjects may or may not be pregnant. There will be no restrictions based on race or ethnic group.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Pressure-induced vasoconstriction of human uterine myometrial arteries [% constriction = ((passive vessel diameter - active vessels diameter) / passive diameter) X 100] | Pressure-induced vasoconstriction will be assessed immediately following specimen acquisition and dissection to isolate the artery of interest. This occurs as a single time point of measurement, less than 24 hours following specimen acquisition.
  Pressure-induced constrictions (PIC) are expressed as a percent decrease of the fully dilated diameter of individual arteries at the same intravascular pressure. Diameter values will be analyzed as percent constriction. The passive diameter of the artery is measured in calcium-free physiologic saline solution containing 80 µM diltiazem. In turn, the active diameter of the myometrial artery is measured in response to calcium-containing physiologic saline solution. Both measurements will be obtained and measured across a physiologic range of blood pressures.

SECONDARY OUTCOMES:
Changes in pressure-induced vasoconstriction in response to blockade of voltage-dependent potassium channels. | Pressure-induced vasoconstriction will be assessed immediately following specimen acquisition and dissection to isolate the artery of interest. This occurs as a single time point of measurement, less than 24 hours following specimen acquisition.
  Pressure-induced constrictions (PIC) are expressed as a percent decrease of the fully dilated diameter of individual arteries at the same intravascular pressure. Diameter values will be analyzed as percent constriction.
Changes in pressure-induced vasoconstriction in response to blockade of prostaglandin production. | Pressure-induced vasoconstriction will be assessed immediately following specimen acquisition and dissection to isolate the artery of interest. This occurs as a single time point of measurement, less than 24 hours following specimen acquisition.
  Pressure-induced constrictions (PIC) are expressed as a percent decrease of the fully dilated diameter of individual arteries at the same intravascular pressure. Diameter values will be analyzed as percent constriction. The passive diameter of the artery is measured in calcium-free physiologic saline solution containing 80 µM diltiazem. In turn, the active diameter of the myometrial artery is measured in response to calcium-containing physiologic saline solution. Both measurements will be obtained and measured across a physiologic range of blood pressures.
Changes in pressure-induced vasoconstriction in response to blockade of nitric oxide synthase. | Pressure-induced vasoconstriction will be assessed immediately following specimen acquisition and dissection to isolate the artery of interest. This occurs as a single time point of measurement, less than 24 hours following specimen acquisition.
  Pressure-induced constrictions (PIC) are expressed as a percent decrease of the fully dilated diameter of individual arteries at the same intravascular pressure. Diameter values will be analyzed as percent constriction. The passive diameter of the artery is measured in calcium-free physiologic saline solution containing 80 µM diltiazem. In turn, the active diameter of the myometrial artery is measured in response to calcium-containing physiologic saline solution. Both measurements will be obtained and measured across a physiologic range of blood pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Leovic, MD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No
Non-applicable